CLINICAL TRIAL: NCT00475618
Title: Effect of Therapeutic Measures in Dental Caries Reduction in Children With Primary Dentition From Metropolitan Area Sorrounded Medellín City. A Clinical Trial
Brief Title: Effect of Therapeutic Measures in Dental Caries Reduction in Children With Primary Dentition From Medellín City
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CES University (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Principal Investigator, Alexandra Saldarriaga Cadavid Ms, Principal investigator, CES University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1-Mejia
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Dental Decay
Keywords: Early chilhood caries; Prevention; Fluoride varnish; fluoride toothpaste; non fluoride tooth paste; Professional cleaning
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluoride Varnish (Experimental): Professional cleaning + education + fluoride vanish
  Interventions: Procedure: topical fluoride varnish application.
- Fluoride Toothpaste 500 ppm (Active Comparator): Professional cleaning + education + fluoride toothpaste 500 ppm
  Interventions: Procedure: professional cleaning
- No fluoride toothpaste (Active Comparator): Professional cleaning + education + no fluoride toothpaste
  Interventions: Procedure: No fluoride toothpaste

INTERVENTIONS:
Procedure: topical fluoride varnish application. — Vanish application every 6 months in all accesible tooth surfaces
  Arms: Fluoride Varnish
Procedure: professional cleaning — Daily use fluoride toothpaste 500 ppm.
  Arms: Fluoride Toothpaste 500 ppm
Procedure: No fluoride toothpaste — Daily use no fluoride toothpaste.
  Arms: No fluoride toothpaste

SUMMARY:
The propouse of this study is to evaluate some combined preventive measures, of easy application in children under 6 years old as education, brush teeth, fluoride free tooth paste,fluoridated tooth paste, professional cleaning and fluoride varnish application, to determine between three groups of differents combined preventive measures, wich one is better in reduting dental caries appearance.

Hypothesis:

1. Ho: Dental caries reduction percentage is larger or equal in the group with only prevention education and Professional cleaning, than in the groups intercepted with fluoride varnish or fluoride toothpaste.
2. Ha: Dental caries reduction percentage is less in the group with only prevention education and Professional cleaning, than in the groups intercepted with fluoride varnish or fluoride toothpaste.

DETAILED DESCRIPTION:
Dental caries is a public health problem in any society. Even though caries prevalence has decreased in many industrialized countries, dental caries in the early infancy still has high prevalence in non developing countries. In Colombia as well Medellín, there are not data of dental caries prevalence in children under 5 years old.

The fact that the official studies do not recognize this world tendency and are limited to age groups over 5 years old, underestimate the disease as an early appearing process in life, specially in underprivileged groups. When dental caries is not properly treated, it becomes a risk factor for other systemic and infectious diseases. Early infant dental caries has been strongly related with malnutrition in children under 6 years old; is has been proved that once their dental problem is treated, weight and size are recovered.

Design and implementation of prevention programs for preschool children must be a priority.This study pretends evaluate some combined preventive measures of easy application in children under 6 as education, brush teeth, fluoride free and fluoridated tooth paste, professional cleaning and fluoride varnish application considering this an easy application measure for this group of age, which eventually it could be more cost-effective than the sealant.

The importance of doing new clinical studies to evaluate the efficacy of fluoride varnishes combined with other preventive measures, is supported in most of other studies have used a non treated group or placebo as a control group.12 The evaluation of the non fluoride toothpaste will give us an exact idea of the contribution of each of the preventive measures in dental caries reduction.

In Colombia, there is not doubt that past preventive programs had a positive effect in dental health of school children. However, preschool children have been out of these programs.

New programs should be carried on to educational establishment and infant care centres without distinction of the type of social health insurance or coverage.

The study pretends to evaluate the efficacy of therapeutics measures like fluoride varnish application and professional cleaning, which are characterized for their low cost and easy application. In the first place, parents and children in the study will receive education lecture, they will be provided with tooth brush and toothpaste with or without fluoride depending the group assigned. At the same time the study pretends to generate knowledge that contributes to minimize invasive and painful treatments in this group of age.

What effect has the inclusion of fluoride varnish and 500 ppm fluoridated toothpaste as preventive measures complementary to oral health education and professional tooth cleaning in reduction of dental caries in children under 5 years old?

Comparisons and Study group design: three groups will be randomly assigned to an experimental group:

1. Group A: Dental health education with brush and 500 PPM fluoride tooth paste; with professional cleaning each 6 months.
2. Group B: Dental health education with brush and non fluoride tooth paste; with professional cleaning each 6 months.
3. Group C: Dental health education with brush and non fluoride tooth paste; with professional cleaning each 6 months and topical fluoride varnish application.

The study will be a random controlled double blind assay made in children with primary dentition and 2.5 or 3.5 years old at the beginning, from socio-economic status 2 and 3 that are attended in Su Salud IPS ( Service lender institution) at the Metropolitan area of Medellín city with 3 years follow-up.

A second part of the study pretends to measure presence of dental fluorosis in the permanent dentition of the children that took part in the first assay. This proposal will be designed in that moment.

ELIGIBILITY:
Inclusion Criteria:

* Children since 2.5 and 3.5 years old
* Deciduous teeth complete formula
* They are part of Su Salud health Service Company
* Healthy chlildrens

Exclusion Criteria:

* children with any mental or fhisical incapacity

Ages: 29 Months to 41 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2007-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Dental Caries reduction as if the patient has or not new dental caries. | Three years with clinical examination every one year.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Saldarriaga, Master of Sience, Principal Investigator — CES University - Medellín - Colombia